CLINICAL TRIAL: NCT00177177
Title: L-Carnosine, an Antioxidant and AGE Inhibitor (Advanced Glycation End Products) for Cognitive Enhancement Among Persons With Schizophrenia: A Randomized, Add-on Double-Blind, Placebo Controlled, Clinical Trial
Brief Title: L-carnosine for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03T-413; IRB #0408179
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: L-carnosine; Schizophrenia; Schizoaffective disorder; Cognitive enhancement
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Carnosine; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): L Carnosine
  Interventions: Drug: L-carnosine (dietary supplement)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: L-carnosine (dietary supplement)

INTERVENTIONS:
Drug: L-carnosine (dietary supplement) — an antioxidant and AGE inhibitor, 500 mg/day, titration each week to reach 2000 mg/day in 4 weeks L-Carnosine is a dietary supplement
  Other Names: L Carnosine; Placebo

SUMMARY:
The investigators' hypothesis is that oral L-carnosine treatment (as compared with placebo) will enhance cognitive abilities (specifically: measures of attention, executive function, working memory, visuospatial ability and language) in persons with schizophrenia or schizoaffective disorder. Secondarily, they hypothesize that there will be secondary improvements in positive, negative and mood symptoms with L-carnosine treatment.

The investigators aim to test these hypotheses by conducting a randomized, placebo controlled, add-on treatment trial of L-carnosine (added to existing antipsychotic treatment) up to 84 recruited subjects with Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) schizophrenia/schizoaffective disorder for a period of 16 weeks. Measures of cognition and psychopathology will be utilized for evaluating primary and secondary outcomes, along with safety assessments.

DETAILED DESCRIPTION:
OBJECTIVE:

Based on the available neuroscience and human data, we hypothesize that supplemental L-carnosine treatment (a potent naturally occuring antioxidant and anti-glycation agent) will be a useful disease modifying agent when used adjunctively with antipsychotic drugs in patients with a diagnosis of either schizophrenia or schizoaffective disorder. More specifically, our hypothesis is that oral L-carnosine treatment (as compared with placebo) will enhance cognitive abilities (specifically: measures of attention, executive function, working memory, visuospatial ability and language) in persons with schizophrenia or schizoaffective disorder. Secondarily, we hypothesize there will be secondary improvements in positive, negative and mood symptoms with L-carnosine treatment.

RESEARCH PLAN:

A randomized, placebo controlled, add-on treatment trial of L-carnosine (added to existing antipsychotic treatment) for a period of 16 weeks. Measures of cognition, and psychopathology will be utilized for evaluating primary and secondary outcomes, along with safety assessments.

METHODS:

Up to eighty-four subjects with DSM-IV-TR schizophrenia/schizoaffective disorder will be recruited from Western Psychiatric Institute and Clinic, Mayview State Hospital, Mon Yough Community Services, Inc. and Dubois Regional Medical Center using a 1:1 randomization, subjects who sign a informed consent document will be randomized to receive L-carnosine or placebo. During a 4 week titration period, the L-carnosine dosage will be increased from 500 to 2000 mg/day, and continued for an additional 8 weeks. If side-effects are noted, a minimum of 500 mg/day of L-carnosine can be used.

A computerized cognitive battery will form the main efficacy measures and be administered at baseline and at visit 6 (i.e. just prior to the 4 week taper); some of these measures will be administered at visit 4 (28 days). Standard psychopathology rating scales will be administered to evaluate secondary aims such as impact on positive and negative symptoms of schizophrenia. Safety will be assessed by tailing a careful medical history and physical examination at screening and evaluating results of laboratory measures. Any adverse effects will be assessed by asking questions at each visit, and if required bringing subjects in for assessments outside the scheduled visits.

SIGNIFICANCE:

Cognitive dysfunction in persons with schizophrenia is a serious limitation to achieving significantly better functional outcomes (Green, et. al., 1996). Till recently, therapeutic nihilism prevailed when it came to treatments that improve cognitive abilities in schizophrenia. One reason for this pessimistic view was that cognitive dysfunction was not considered to be malleable to treatment but instead was thought to represent an unchanging dimension of the illness. However, that view is now changing, and psychosocial and cognitive remediation techniques are being evaluated to treat cognitive dysfunction in schizophrenia. A recent synthesis of data would suggest that mediators of a better cognitive outcome may also include agents that target the inefficient antioxidant defenses in persons with schizophrenia, or those that counter NMDA-glutamate neuronal excitotoxicity (Yao et al., 2001). These mechanisms may underlie the neuronal membrane pathology in schizophrenia, and in turn these abnormalities may contribute to the cognitive dysfunction and decline reported during the course of the illness. The benefits of L-carnosine (a naturally occurring antioxidant and anti-glycation agent) for improved cognitive abilities and in social behavior and communicative skills were reported in a random-assignment, double-blind, placebo-controlled trial in children and adolescents with autism; specifically improvements in receptive language scores and socialization and communication skill scores (Chez et al., 2002a).

The primary focus of this study is to evaluate the ability of L-carnosine, a naturally occurring dipeptide, to enhance cognitive abilities in people with schizophrenia. The study will also evaluate whether L-carnosine has secondary benefits for positive and negative and mood symptoms. As a relatively benign agent, L-carnosine offers the potential to achieve a significant clinical impact in improving cognitive dysfunction in persons with schizophrenia, if efficacy is confirmed.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR diagnosis of schizophrenia (any subtype, except currently catatonic) or schizoaffective disorder
* Ages 18 to 65 years
* Men or women
* Ability to read and communicate in English
* 8th grade education or greater
* Ability to provide informed, competent and written consent
* Current antipsychotic medication is stable for greater than or equal to 4 weeks.

Exclusion Criteria:

* Medically unstable conditions
* Known allergy to L-carnosine
* Current cognitive decline is attributable to a diagnosis of dementia or other neurological disorder
* Pregnant or lactating women
* Mini-mental state examination score (MMSE) less than or equal to 23
* HIV positive status resulting in AIDS-related dementia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To see if oral L-carnosine treatment (as compared with placebo) will enhance cognitive abilities (as noted below) | 12 weeks treatment
executive function, working memory, attention, visuospatial ability | 12 weeks treatment

SECONDARY OUTCOMES:
To examine if secondary improvements in positive, negative and mood symptoms occur with L-carnosine treatment | 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: K.N. Roy Chengappa, MD, Principal Investigator — Western Psychiatric Institute and Clinic
Locations (4):
- United States (4):
  - Mayview State Hospital, Bridgeville, Pennsylvania
  - Dubois Regional Medical Center, DuBois, Pennsylvania
  - Mon-Yough Community Services, Inc., McKeesport, Pennsylvania
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Chengappa KN, Turkin SR, DeSanti S, Bowie CR, Brar JS, Schlicht PJ, Murphy SL, Hetrick ML, Bilder R, Fleet D. A preliminary, randomized, double-blind, placebo-controlled trial of L-carnosine to improve cognition in schizophrenia. Schizophr Res. 2012 Dec;142(1-3):145-52. doi: 10.1016/j.schres.2012.10.001. Epub 2012 Oct 23. PMID 23099060